CLINICAL TRIAL: NCT05715099
Title: Efficacy of Nutritional Saffron Supplement as an Anti-inflammatory Agent in Egyptian Patients With Inflammatory Bowel Disease
Brief Title: Saffron as Anti Inflammatory In Patients With Inflammatory Bowel Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Alshymaa Hassnine, associated prof, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SaffronIBD
Record Dates: First submitted 2023-01-19; First posted 2023-02-06 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — safranal

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- mild-moderate ulcerative colitis for low dose (Active Comparator): 2 low dose (25 mg \dose) per day N= 20
  Interventions: Drug: Saffron
- mild-moderate ulcerative colitis for high dose (Active Comparator): 2 high dose (50 mg \dose) per day N=20
  Interventions: Drug: Saffron
- healthy subjects for low dose (Active Comparator): 2 low dose (25 mg \dose) per day N= 10
  Interventions: Drug: Saffron
- healthy subjects for high dose (Active Comparator): 2 high dose (50 mg \dose) per day N=10
  Interventions: Drug: Saffron
- mild-moderate ulcerative colitis for placebo (Placebo Comparator): 2 dose placebo per day N=20
  Interventions: Drug: Placebo
- healthy subjects for placebo (Placebo Comparator): 2 dose placebo per day N=10
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Saffron — Dietary Supplement: saffron supplement for IBD
  Other Names: safranal
  Arms: healthy subjects for high dose; healthy subjects for low dose; mild-moderate ulcerative colitis for high dose; mild-moderate ulcerative colitis for low dose
Drug: Placebo — Dietary Supplement: placebo for IBD
  Arms: healthy subjects for placebo; mild-moderate ulcerative colitis for placebo

SUMMARY:
Nutritional Saffron supplement has been widely used as food supplement and has known anti-depressant and anti-inflammatory activities. The investigators use saffron extract in Egyptian patients with ulcerative colitis for 8 weeks.

DETAILED DESCRIPTION:
The patients invited to participate in a research study on Inflammatory Bowel Diseases (IBD) and saffron as a nutritional anti-inflammatory supplement.

Inflammatory Bowel Disease (IBD) is composed of Crohn's Disease (CD) and Ulcerative Colitis (UC). Continuous altered immune responses and inflammation associate with this disease. More than two-thirds of patients reported that IBD-associated symptoms negatively affected their quality of life and their performance at work.

* Patients with IBD are generally put on immunosuppressants (that block or slow participants' immune system to lower the level of inflammation). Long-term use of these immunosuppressants have some serious side effects.
* The goal of this protocol is to lower the need for these immunosuppressants by giving saffron as capsules in two different doses. The investigators will assess whether the addition of saffron will improve the overall patient's status and decrease the need for immunosuppressants. If participants have been prescribed immunosuppressants by the participant's doctor, saffron will be added to the participants' treatment.
* The investigators request that the subject answer as many questions as they can during this visit. If they are unable to complete the questionnaires during this visit, the investigators ask them to please return them within 7 days. If the investigators do not receive the questionnaires, the investigators will make one phone call to remind the subjects to send the questionnaires back.
* The subject medical record and colonoscopy report will be used to determine IBD or health status, the blood sample will be used to assess immune markers (inflammatory and antiinflammatory), stool sample will be used to assess some inflammation markers and saffron effect on the intestinal bacterial composition, a saliva sample will be used to assess whether saffron selectively affects the intestinal bacteria but not the saliva bacteria and the urine sample will be used to assess saffron release in body fluids.
* Participants are being asked to participate in this research project because participants are having a normal colonoscopy for screening, or IBD.
* If a biopsy is taken at colonoscopy. a pathologist will use a portion to make a diagnosis. The investigators are requesting permission to use a portion of the excess tissue that the pathologist does not need, for this research project.
* Samples will be collected at baseline (day 0) and 8 weeks later after saffron capsules utilization.
* This is a double-blind clinical trial, you will not know whether participants are given a placebo (capsule without saffron) or saffron dose 1 or 2. This is important for participants and for the study process, to avoid any psychological effect on the expected saffron effect.
* However, by the end of the 8 weeks and after collecting and analyzing the data from all participants, the investigators will inform the subject of what the subjects were given and potential next steps.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged >18 years
2. Have UC diagnosed at least 3 months prior to screening? The diagnosis of UC must be confirmed by endoscopic and histologic evidence.
3. Men and women of childbearing potential must agree to use adequate birth control measures during the study.
4. Ability to provide written informed consent and to be compliant with the schedule of protocol assessments, treatment plan, laboratory tests, and other study procedures.
5. UC patients with mild, mod, severity as assess by the 4 scale assessment (Normal, mild, mod, severe).
6. Treatment naïve subjects diagnosed with ulcerative colitis (without previous exposure to treatment).

7. UC patients already on a treatment might be considered, with saffron as an add-on 8. UC patients who displayed no improvement with any available treatment might be considered for saffron as an alternative treatment in this option.

Exclusion Criteria:

* 1 Patients taking immunosuppressive medicine for a disease other than UC 2 Rheumatologic disease and other underlying diseases that can interfere with the study process.

  3 Pregnancy 4 If the UC has been present for > 10 years, a colonoscopy with biopsy has to be performed to rule-out dysplasia.

  5 A subject who had surgery as a treatment for ulcerative colitis or likely to require surgery during the study period.

  6 Subjects with evidence of liver disease or abnormal liver enzymes and function tests (e.g. total bilirubin, aspartate aminotransferase (AST) or alanine aminotransferase (ALT) higher than the upper limit of normal) at the screening visit.

  7 Subjects who have any condition possibly affecting oral nutritional supplement absorption.

  8 Any other condition which in the opinion of the investigators would make the subject unsuitable for inclusion in the study.

  9 Patients with known active or untreated GI infections including C. difficile, CMV, HSV, HIV

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-03-30 (Estimated); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
fecal calprotectin assessment | 8 weeks
  Decrease in calprotectin levels. Fecal calprotectin normal range to be 10 to 60 μg/mg
C reactive protein assessment | 8 weeks
  change on C reactive protein level reading is less than 10 milligram per liter
erythrocyte sedimentation rate assessment | 8 weeks
  maintaining erythrocyte sedimentation rate with the normal range of 0 to 22 mm/hr for men and 0 to 29 mm/hr for women
The Ulcerative Colitis Colonoscopic Index of Severity scores | 8 weeks
  Decrease of 2 or more unit in the Ulcerative Colitis Colonoscopic Index of Severity score. The Ulcerative Colitis Colonoscopic Index of Severity scores for mild colitis is 3-5, and for moderate is 5-9

SECONDARY OUTCOMES:
endoscopy colitis assessment | 8-12 weeks
  Secondary endpoints will be endoscopy remission at week 8-12 according to gastroenterologist preference

CONTACTS AND LOCATIONS:
Locations (1):
- Minia University, Minya, Minya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No